CLINICAL TRIAL: NCT05947097
Title: An Open-label, Single-dose Study to Assess the Pharmacokinetics of HSK21542 Injection in Subjects With Varying Degrees of Renal Impairment Compared to the Control Subjects With Normal Renal Function
Brief Title: A Study to Evaluate the Pharmacokinetics of HSK21542 in Subjects With Renal Impairment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK21542-104
Record Dates: First submitted 2023-06-29; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mild Renal Impairment (Experimental)
  Interventions: Drug: HSK21542 Injection
- Moderate Renal Impairment (Experimental)
  Interventions: Drug: HSK21542 Injection
- Severe Renal Impairment (Experimental)
  Interventions: Drug: HSK21542 Injection
- Normal Renal function (Experimental)
  Interventions: Drug: HSK21542 Injection

INTERVENTIONS:
Drug: HSK21542 Injection — 1ug/kg bolus for 2min±5s

SUMMARY:
This is an open-label, single-dose study to evaluate the pharmacokinetics and safety of HSK21542 in subjects with mild, moderate and severe renal impairment compared to the matched control subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

Subjects with renal impairment(RI):

1. Voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions;
2. 18 years to 79 years (inclusive), male and female;
3. Male subjects weight ≥50 kg and female subjects weight ≥45 kg. Body mass index (BMI) : 18-30 kg/m2 (inclusive) (BMI= weight (kg)/height2 (m^2));
4. Subjects with medically stable RI until study completion corresponding to the classifications of Renal Function based on GFR: mild RI: 60≤GFR<90 mL/min; moderate RI: 30≤GFR<60 mL/min, severe RI:15≤GFR<30 mL/min;
5. Physical examination, vital sign measurements, 12-lead electrocardiogram (ECG), and clinical laboratory tests results were deemed appropriate by the investigator;
6. Not in use of any drug within 2 weeks prior to screening, except for the medication necessary for RI/ other comorbidities (last more than four weeks in good compliance);
7. Subjects (including partners) are willing to voluntarily use effective contraceptives from screening to at least 6 months after the last dose administration.

Subjects with normal renal function :

1. Voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions;
2. 18 years to 79 years (inclusive), male and female, age and sex must be matched with subjects with RI;
3. Male subjects weight ≥50 kg and female subjects weight ≥45 kg, weight must be matched with subjects with RI. Body mass index (BMI) : 18-30 kg/m^2 (inclusive) (BMI= weight (kg)/height2 (m^2));
4. 90≤GFR<130 mL/min;
5. Physical examination, vital sign measurements, 12-lead electrocardiogram (ECG), and clinical laboratory tests results were deemed appropriate by the investigator;
6. Not in use of any drug within 2 weeks prior to screening, except for the medication necessary for comorbidities (last more than four weeks in good compliance);
7. Subjects (including partners) are willing to voluntarily use effective contraceptives from screening to at least 6 months after the last dose administration.

Exclusion Criteria:

1. Subjects who have a allergic to any component of HSK21542 injection or allergic history to opiates, such as urticaria (opiate-related adverse reactions such as constipation and nausea are not included as exclusion criteria in this study);
2. Have a history of severe and uncontrolled diseases, such as cardiovascular, respiratory, liver, gastrointestinal, endocrine, hematologic, mental/nervous systems diseases within one year prior to screening;
3. Have conditions that may affect drug absorption, distribution, metabolism, or excretion (e.g., disease, drugs or surgery);
4. Acute renal failure;
5. Smoking more than 5 cigarettes per day within 3 months prior to screening or smoking during the study;
6. Average alcohol intake is more than 14 unit per week (1unit=17.7 mL alcohol , 1 unit=357mL 5% alcohol beer, or 43mL 40% alcohol spirit, or 147mL 12% alcohol wine) within the 3 months prior to screening, or taking any alcohol during study or a positive ethanol breath test at screening;
7. Drug abuse history within 5 years prior to screening, or positive urine drug screen at screening;
8. History of high consumption of grapefruit juice, methylxanthine-rich food or beverage (such as coffee, tea, cola, chocolate, energy drinks) ,consumption of grapefruit juice, methylxanthine-rich food within 48 hours before the administration;
9. Participation in another clinical trial within 3 months before screening;
10. Blood donation (or blood loss) ≥400 mL, or receiving blood products to improve anemia within 3 months prior to the screening;
11. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 2 × upper limit of normal, or bilirubin > 1.5 × upper limit of normal;
12. Have a positive result for hepatitis B surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, or anti-treponema pallidum specific antibody;
13. A pregnant/lactating woman, or has a positive pregnancy test at screening or during the trial;
14. Not suitable for this study as judged by the investigator.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | From the start to 240 hours after bolus
  The maximun plasma concentration of HSK21542
AUC0-t | From the start to 240 hours after bolus
  Area under the concentration-time curve from time zero to time of last quantifiable concentration
AUC0-inf | From the start to 240 hours after bolus
  Area under the concentration-time curve from time zero extrapolated to infinite time

SECONDARY OUTCOMES:
Tmax | From the start to 240 hours after bolus
  Time of maximum concentration
t1/2 | From the start to 240 hours after bolus
  half-life
Vz | From the start to 240 hours after bolus
  Volume of distribution associated with the terminal phase
CL | From the start to 240 hours after bolus
  Plasma clearance
Ae | Predose and 72 hours after dosing
  Cumulative urinary recovery of unchanged drug
Fe | Predose and 72 hours after dosing
  Cumulative urinary recovery fraction of unchanged drug
CLr | Predose and 72 hours after dosing
  Renal clearance

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, PhD, Principal Investigator — Qianfoshan Hospital
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No